CLINICAL TRIAL: NCT04248920
Title: Clinic to Community© Program for Adults With Epilepsy Admitted to Emergency Departments: A Randomized Controlled Trial
Brief Title: Clinic to Community© Program for Adults With Epilepsy Admitted to Emergency Departments
Acronym: C2CEDRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Ontario Brain Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 9045
Record Dates: First submitted 2020-01-15; First posted 2020-01-30 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Epilepsy, Generalized
Keywords: Health Care Utilization; Emergency Department
MeSH Terms: conditions — Epilepsy, Generalized; Patient Acceptance of Health Care; Emergencies

STUDY DESIGN:
Intervention Model Description: This is a parallel, pilot randomized controlled trial (RCT) comparing the Clinic To Community© program plus treatment-as-usual (TAU) with TAU only (i.e. wait-list control).
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, it is not feasible for participants and study personnel to be blinded. However, the letter of information (LOI) indicates that the study aims to evaluate outcomes after an ED visit, and, in addition, evaluate the impact of a community engagement program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention Group. Participants randomized to the intervention group will complete the C2C program. They will receive an in-person one-on-one 60-minute education session and will be introduced to, and encouraged to participate in, the programs and support services that are provided by Epilepsy Southwestern Ontario (ESWO). As part of the C2C program, participants will be contacted 6 months later for a supplementary consultation over the telephone and to answer any questions. Epilepsy is unique among chronic, episodic disorders in that PWE lose their ability to make choices during a seizure and depend to a greater degree on the decisions of others including family, friends and colleagues. For this reason, we encourage the PWE to invite their support network to attend the patient education sessions.
  Interventions: Behavioral: Clinic to Community Education Program
- Waitlist Control Group (Other): Waitlist Control Group. The control group continues TAU and will be followed up 12 months after randomization. The control group will receive C2C after the 12-month follow-up.
  Interventions: Behavioral: Clinic to Community Education Program

INTERVENTIONS:
Behavioral: Clinic to Community Education Program — The C2C program aims to improve participants' knowledge of epilepsy and access to services and to provide support. Participants randomized to the intervention group will complete the C2C program. They will receive an in-person one-on-one 60-minute education session and will be introduced to, and encouraged to participate in, the programs and support services that are provided by Epilepsy Southwestern Ontario (ESWO).

SUMMARY:
Analysis of emergency department (ED) visits with a billing code for 'epilepsy' or 'seizure' found up to 37% are eligible for deferral. This study is a randomized controlled trial (RCT) of the Clinic To Community© program (C2C) as an intervention for adults with epilepsy visiting emergency departments at a mid size hospital in Ontario, Canada. Participants in the intervention arm receive patient education to improve knowledge of epilepsy and access to community-based services. Participants in the control group are wait-listed and receive patient education 12 months later. The study objective is to successfully implement, recruit and retain participants for this intervention and evaluate whether C2C will reduce the frequency of ED visits, reduce felt stigma and improve quality of life, epilepsy knowledge, and self-management skills.

DETAILED DESCRIPTION:
Emergency care for epilepsy can be appropriate and even life-saving, but up to 37% of emergency department (ED) visits by persons with epilepsy (PWE) are potentially deferrable, resulting from persons with known epilepsy and uncomplicated seizures. Past studies have shown that low self-management confidence among PWE leads to frequent emergency visits to the hospital. Other factors associated with increased use of EDs are increased seizure frequency, reduced medication, sub-optimal self-management, increased anxiety, increased depression, increased felt-stigma, and lower social and medical epilepsy knowledge.

In one catchment area in Ontario, Canada, the Southwest Local Health Integration Network (LHIN), there are an estimated 7508 prevalent cases of epilepsy associated with the use of approximately $55 million/year of provincial healthcare services. In addition, there are an estimated 433 incident cases costing an additional $4.6 million/year. Hospital care (including ED visits) accounts for 35.5% of the total cost equating to $21 million/year. Eliminating the 37% of deferrable ED visits equates to saving almost $8 million/year.

The Clinic to Community© (C2C) epilepsy education program has been developed using best practices for patient education. The content has been divided into an introductory 60 minute face-to-face session supported by strategy sheets that can be accessed online at www.clinictocommunity.ca

The Clinic To Community© program recognizes that epilepsy is unique among chronic conditions in that PWE lose their ability to make choices during a seizure and depend on the decisions of others including family, friends and colleagues to keep them safe. Many patients seek care in the ED to reduce their anxiety and for reassurance and that upon discharge from the ED, the inability to receive a prompt specialist appointment leads to the continued use of ED for these same patients.

This is a parallel, pilot randomized controlled trial (RCT) comparing the Clinic To Community© program plus treatment-as-usual (TAU) with TAU only (i.e. wait-list control). This study will not interfere with patients' clinical care. Eligible patients visiting a participating ED will be given information about the study and if they agree, will be referred. The C2C program will be delivered in-person, one-on-one for 60 minutes by appointment on a rolling basis to minimize wait-times and allow timely access to the intervention.

All participants will complete questionnaires before randomization and 12 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (aged ≥18 years) visiting a participating ED for a seizure or an epilepsy-related concern.
2. Adults on anti-seizure medication prior to coming to the ED or prescribed anti-seizure medication at the ED.
3. Providing informed consent and having sufficient English language skills to complete questionnaires and participate in the intervention.

Exclusion Criteria:

1. Previous participation in the C2C program.
2. Known diagnosis of psychogenic non-epileptic seizures (PNES).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Rate of engagement with the Clinic To Community© (C2C) program | Throughout study completion, approximately 2 years
  Evaluated by rate of ED referrals, rate of recruitment, rate of retention, and proportion who receive support education.

SECONDARY OUTCOMES:
Frequency of epilepsy-related emergency department (ED) visits over the next 12 months | Baseline (0), and 12 months
  Change from baseline in frequency of ED visits and health care utilization, adapted from the Canadian Community Health Survey
Effect of participation in C2C on felt stigma using "Stigma Scale of Epilepsy" | Baseline (0) and 12 months
  Change from baseline in using the Stigma Scale of Epilepsy, 3-item scale asking: "Because of epilepsy, (1) other people are uncomfortable with me; (2) treat me as inferior; (3) prefer to avoid me." Each of those questions is scored on a four-point scale:
  0 not at all; 1 yes, maybe; 2 yes, probably; 3 yes, definitely. Total scores range from 0 to 9 and categorized as not stigmatized (score of 0), mild-moderate (1-6) and highly stigmatized (7-9).
Effect of participation in C2C on felt stigma using "Epilepsy Stigma Scale" | Baseline (0) and 12 months
  Change from baseline measured by Epilepsy Stigma Scale, a 10-item measure evaluating stigma. Items are measured on a 7-point Likert Scale, from "strongly agree" to "strongly disagree".
Effect of participation in C2C on self-management skills | Baseline (0) and 12 months
  Change from baseline measured by the Adult Epilepsy Self-Management Measurement Instrument (AESMMI-65) This measure is a 65-item scale assessing the frequency of use of epilepsy self-management practises. Contains seven domains: 1) healthcare communication, 2) treatment management, 3) coping, 4) social support, 5) seizure tracking, 6) wellness, and 7) seizure response.
Effect of participation in C2C on quality of life | Baseline (0) and 12 months
  Change from baseline measured by Quality of Life in Epilepsy Inventory (QOLIE 10), a 10-item scaled evaluating quality of life in adults with epilepsy. Responses range from "all of the time" to "none of the time"
Effect of participation in C2C on epilepsy knowledge | Baseline (0) and 12 months
  Change from baseline on the "Thinking About Epilepsy Questionnaire" knowledge subscale. Knowledge is assessed by answering true/false/I don't know

OTHER OUTCOMES:
Effect on quality of life using World Health Organization Quality of Life (WHOQOL) | Baseline (0) and 12 months
  Change from baseline measured by World Health Organization Quality of Life (WHOQOL) - Abbreviated (BREF), 30-item measure of quality of life, generic-HRQOL instrument.
Effect on activities of daily living using Sheehan Disability Scale | Baseline (0) and 12 months
  Change from baseline measured by the Sheehan Disability Scale is 5-items for patient-rated measure of disability and impairment.
Effect on anxiety using Generalized Anxiety Disorder 7-item (GAD-7) scale | Baseline (0) and 12 months
  Change from baseline using the Generalized Anxiety Disorder 7-item (GAD-7) scale, 7-item scale evaluating generalized anxiety. Generates an overall anxiety score, with scores above 10 indicative of moderate-severe anxiety.
Effect on depressive symptoms based on Quick Inventory of Depressive Symptomatology | Baseline (0) and 12 months
  Change from baseline using the Quick Inventory of Depressive Symptomatology, 14-item scale evaluating depressive symptoms.
Effect on sleep quality using Pittsburgh Sleep Quality Index (25-items) | Baseline (0) and 12 months
  Change from baseline measured by the Pittsburgh Sleep Quality Index, 25-item scale evaluating sleep quality.
Effect on suicide ideation using Columbia-Suicide Severity Rating Scale (C-SSRS) Screener | Baseline (0) and 12 months
  Change from baseline measured by the C-SSRS Screener, a 6-item scale evaluating suicidal ideation.
Effect on Psychiatric comorbidities using Brief Symptom Inventory | Baseline (0) and 12 months
  Change from baseline measured by 53-items covering nine symptom dimensions: Somatization, Obsession-Compulsion, Interpersonal Sensitivity, Depression, Anxiety, Hostility, Phobic anxiety, Paranoid ideation and Psychoticism; and three global indices of distress: Global Severity Index, Positive Symptom Distress Index, and Positive Symptom Total. The global indices measure current or past level of symptomatology, intensity of symptoms, and number of reported symptoms, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Kathy N Speechley, PhD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
This study is partnered with the Ontario Brain Institute (OBI). Study data and other personal health information collected as a part of this research study will be shared with the Ontario Brain Institute. OBI is a not-for profit research institute that funds people to work together to find cures and better treatments for brain disorders. It includes not just doctors and researchers but patients, members of the medical community, government and other health-related organizations. This database of research data is known as 'Brain-CODE'.
  Brain-CODE is an open-access database. This means that researchers and organizations outside of this study can request access to study data that is in the Brain-CODE database. OBI may take data, combine it with data from many other people, and make it available to enhance the public's awareness of research. They will use tools to remove identifying information from these combined data sets, making the risk of identifiers minimal.
Supporting Information: SAP, ICF
Time Frame: Data will be stored in BrainCODE indefinitely
Access Criteria: Access to data by outside researchers or organizations will require a detailed plan for the use of the data, and approval from a research ethics board, as described in OBI's Data Sharing Policy http://www.braininstitute.ca/Brain-CODE-governance. These researchers or organizations will be required to enter into an agreement with OBI that clearly states the safeguards that will be in place to protect that data, and the purposes for which this data may be collected, used, stored and disclosed.
URL: http://www.braininstitute.ca/Brain-CODE-governance

REFERENCES:
- [Background] Bautista RE, Glen ET, Wludyka PS, Shetty NK. Factors associated with utilization of healthcare resources among epilepsy patients. Epilepsy Res. 2008 May;79(2-3):120-9. doi: 10.1016/j.eplepsyres.2008.01.003. Epub 2008 Mar 12. PMID 18339521
- [Background] Bowen JM, Snead OC, Chandra K, Blackhouse G, Goeree R. Epilepsy care in ontario: an economic analysis of increasing access to epilepsy surgery. Ont Health Technol Assess Ser. 2012;12(18):1-41. Epub 2012 Jul 1. PMID 23074428
- [Background] Couldridge L, Kendall S, March A. A systematic overview--a decade of research'. The information and counselling needs of people with epilepsy. Seizure. 2001 Dec;10(8):605-14. doi: 10.1053/seiz.2001.0652. PMID 11792167
- [Background] Noble AJ, Mathieson A, Ridsdale L, Holmes EA, Morgan M, McKinlay A, Dickson JM, Jackson M, Hughes DA, Goodacre S, Marson AG. Developing patient-centred, feasible alternative care for adult emergency department users with epilepsy: protocol for the mixed-methods observational 'Collaborate' project. BMJ Open. 2019 Nov 2;9(11):e031696. doi: 10.1136/bmjopen-2019-031696. PMID 31678950
- [Background] Kapoor, Deepa, Joubert, Gary, Thind, Amardeep, Secco, Mary, Speechley, Kathy Nixon. Number of Potentially Deferrable Patients Presenting to Emergency Departments in London with Seizures. Epilepsia 2007; Vol 48, Supplement 6